CLINICAL TRIAL: NCT05394493
Title: An Observational Chart Review Study to Describe the Real-world Outcomes and Use of Avelumab in Combination With Axitinib for Treatment of Patients With Advanced Renal Cell Carcinoma in the United Kingdom.
Brief Title: An Observational Chart Review Study To Describe The Real-World Outcomes And Use Of Avelumab In Combination With Axitinib For Treatment Of Patients With aRCC In The UK
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B9991044
Record Dates: First submitted 2022-05-23; First posted 2022-05-27 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Advanced Renal Cell Carcinoma
MeSH Terms: interventions — avelumab; Axitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- patients with advanced renal cell carcinoma
  Interventions: Drug: avelumab; Drug: axitinib

INTERVENTIONS:
Drug: avelumab — as provided in real world setting
Drug: axitinib — as provided in real world settings

SUMMARY:
An observational chart review study to describe the real-world outcomes and use of avelumab in combination with axitinib for treatment of patients with advanced renal cell carcinoma in the United Kingdom.

ELIGIBILITY:
Inclusion criteria

* Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:
* Patients with a documented diagnosis of aRCC.
* Patients aged ≥18 years old at the index event date.
* Patient initiated on treatment with avelumab in combination with axitinib ( ≥1 dose) on or after 1st August 2019.

Exclusion criteria

* Patients meeting any of the following criteria will not be included in the study:
* Patients who received avelumab in combination with axitinib as part of a clinical trial
* Patients initiated on avelumab in combination with axitinib less than 12 months from the end of data collection.
* Patients who are known to have opted out of participation in any research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in between 10 and 15 National Health Service (NHS) hospital trusts and Health Boards
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Objective response (OR) | August 2019 through July 2023
  "Percentage of participants with objective response based assessment of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST).
  CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short aixs was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
  "
Overall Survival (OS) | August 2019 through July 2023
  Time in weeks or months from randomization (or the start of study treatment for non-randomized studies) to date of death due to any cause. OS was calculated as (the death date or last known alive date (if death date unavailable) minus the date of randomization (or first dose of study medication for non-randomized studies) plus 1) divided by 7 or 30.44 if in months.
Progression Free Survival (PFS) | August 2019 through July 2023
  Median time from the first dose of study treatment to the first documentation of objective tumor progression or to death due to any cause, whichever occurs first. PFS calculated as (Weeks) = (first event date minus first dose date plus 1) divided by 7
Duration of Response (DoR) | August 2019 through July 2023
  Median duration (50%) of tumor response for a subgroup of participants with objective disease response: who have not progressed or died due to any cause; with a response and subsequent progression or death due to any cause for DR. DR defined as time from start of first documented objective tumor response [Complete Response (CR) or Partial Response (PR)] to first documented objective tumor progression or death due to any cause, whichever occurs first. DR calculated as (Weeks) = (the end date for DR minus first subsequent confirmed CR or PR plus 1) divided by 7.
Duration of Treatment (DoT) | August 2019 through July 2023

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Ltd, Sandwich, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Ged Y, Markowski MC, Singla N, Rowe SP. The shifting treatment paradigm of metastatic renal cell carcinoma. Nat Rev Urol. 2022 Nov;19(11):631-632. doi: 10.1038/s41585-022-00651-9. PMID 36064785
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B9991044